CLINICAL TRIAL: NCT01516359
Title: Official Title is Required by the WHO and ICMJE
Brief Title: Incidence and Predictive Factors of Intestinal Injury in Patients Undergoing Heart Valve Replacements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cai Li (Other)
Responsible Party: Sponsor-Investigator, Cai Li, Vice head of Dept. of Anesthesiology, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: intestinal injury
Record Dates: First submitted 2012-01-16; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Injury of Other and Multiple Parts of Small Intestine

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are retained for the detections of some biomarkers and gene polymorphism.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with cardiac surgery

SUMMARY:
The purpose of this study is to investigate the incidence and predictive factors related to intestinal injury in patients undergoing heart valve replacement through a multicenter study in China.

DETAILED DESCRIPTION:
Intestinal injury is one of main reasons for mobidity and mortality after heart valve replacement, but its incidence and potential risk factors remain unclear. A multicenter study in China is undertaken to investigate the incidence and predictive factors related to intestinal injury in patients undergoing heart valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing heart valve replacements under cardiopulmonary bypass

Exclusion Criteria:

* Patients who die during or after operation

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing heart valve replacements under cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
score of gut dysfunction | eight months
  At different time points, gut dysfunction is graded according to previous criterion.

SECONDARY OUTCOMES:
The duration of cardiopulmonary bypass | Eight months
  Record the duration of cardiopulmonary bypass
The duration for aortic artery clamping | eight months

CONTACTS AND LOCATIONS:
Overall Officials: Ke Xuan Liu, MD, Ph.D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Anesthesiology, The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China